CLINICAL TRIAL: NCT00320190
Title: An Open-label, Randomized Study of Dasatinib vs High-dose (800-mg) Imatinib in the Treatment of Subjects With Chronic Phase Chronic Myeloid Leukemia Who Have Had a Suboptimal Response After at Least 3 Months of Therapy With 400 mg Imatinib
Brief Title: Study of Dasatinib in Patients With Chronic Phase Chronic Myeloid Leukemia and a Suboptimal Response to Imatinib
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Terminated due to slow participant accrual
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA180-043; EUDRACT Number: 2005-005153-22
Record Dates: First submitted 2006-05-01; First posted 2006-05-03 (Estimated); Results first posted 2011-07-07 (Estimated); Last update posted 2013-10-30 (Estimated); Status verified 2011-07

CONDITIONS: Leukemia, Myeloid, Chronic
Keywords: Chronic phase CML, with a suboptimal response after treatment with imatinib
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Leukemia, Myeloid, Chronic-Phase | interventions — Imatinib Mesylate; Dasatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dasatinib (Active Comparator): Participants with chronic phase chronic myeloid leukemia (CML) who had only a suboptimal response after at least 3 months of therapy with imatinib, 400 mg.
  Interventions: Drug: Dasatinib
- Imatinib (Active Comparator): Participants with chronic phase CML who had only a suboptimal response after at least 3 months of therapy with imatinib, 400 mg.
  Interventions: Drug: Imatinib

INTERVENTIONS:
Drug: Imatinib — Imatinib tablets administered orally at a dose of 400 mg twice daily. Each 400- mg dose to be taken with a meal and a large glass of water.
  Arms: Imatinib
Drug: Dasatinib — Dasatinib tablets administered orally at a dose of 100 mg once daily.
  Arms: Dasatinib

SUMMARY:
The purpose of this study is to compare the efficacy of dasatinib with that of high-dose (800-mg) imatinib in participants with chronic phase chronic myeloid leukemia who achieved only a suboptimal response after at least 3 months of monotherapy with 400-mg imatinib. The safety of these treatments will also be evaluated.

DETAILED DESCRIPTION:
Participants were randomized 2:1 to dasatinib or high-dose imatinib, respectively. Randomization was stratified by a suboptimal response, defined as a hematologic response less than a complete hematologic response after at least 3 months of monotherapy with 400-mg imatinib; a cytogenic response (CgR) less than a partial CgR (PCgR) after at least 6 months of monotherapy with 400-mg; a PCgR after at least 12 months of monotherapy with 400-mg imatinib; or less than a major molecular response with a complete CgR after at least 18 months of monotherapy with 400-mg imatinib.

Participants received either dasatinib or imatinib for 12 months or until disease progression, unacceptable toxicity, consent withdrawal, or study discontinuation. After 12 months, who had a confirmed major molecular response and were still receiving dasatinib, 100 mg, or imatinib, 800 mg, were eligible to extend treatment for an additional 12 months. Participants permanently discontinuing treatment before 12 months were considered treatment failures and withdrawn from the study.

ELIGIBILITY:
Inclusion Criteria:

* Chronic phase Ph^+ chronic myeloid leukemia (CML) demonstrating only a suboptimal response, defined as a hematologic response that is less than a complete hematologic response after at least 3 months of monotherapy with imatinib, 400 mg; a cytogenic response (CgR) that is less than a partial CgR (PCgR) after at least 6 months of monotherapy with imatinib, 400 mg; a PCgR after at least 12 months of monotherapy with imatinib, 400 mg; or less than a major molecular response with a complete CgR after at least 18 months of monotherapy with imatinib, 400 mg.
* Either gender
* Age of 18 years or older

Exclusion Criteria:

* Previous diagnosis of accelerated phase or blast crisis CML
* Uncontrolled or significant cardiovascular disease
* History of significant bleeding disorder unrelated to CML
* Concurrent malignancies
* Intolerance of imatinib, 400 mg
* Prior treatment with imatinib at a dose higher than 400 mg
* Prior stem cell transplantation and/or high-dose chemotherapy for CML

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2006-08; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (25):
- Belgium (2):
  - Local Institution, Antwerp
  - Local Institution, Charleroi
- Finland (2):
  - Local Institution, Helsinki
  - Local Institution, Tampere
- France (7):
  - Local Institution, Lyon
  - Local Institution, Marseille
  - Local Institution, Montpellier
  - Local Institution, Paris
  - Local Institution, Rennes
  - Local Institution, Strasbourg
  - Local Institution, Toulouse
- Local Institution, Leipzig, Germany
- Local Institution, Orbassano (To), Italy
- Norway (2):
  - Local Institution, Oslo
  - Local Institution, Trondheim
- Local Institution, Lisbon, Portugal
- Russia (2):
  - Local Institution, Moscow
  - Local Institution, Saint Petersburg
- Local Institution, Murcia, Spain
- Sweden (3):
  - Local Institution, Lund
  - Local Institution, Örebro
  - Local Institution, Uppsala
- United Kingdom (3):
  - Local Institution, Glasgow, Central
  - Local Institution, London, Greater London
  - Local Institution, Leeds, North Yorkshire

REFERENCES:
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of 52 participants enrolled, 32 were randomized to treatment. Of the 20 not randomized, 17 no longer met study criteria, 1 participant had an adverse event prior to randomization, 1 participant was enrolled after the sponsor stopped recruitment, and 1 participant was stopped due to administrative reasons.
Groups:
- Dasatinib, 100 mg: Dasatinib, 100 mg, administered orally once daily.
- Imatinib, 800 mg: Imatinib, 400 mg, administered orally twice daily.
Period: First 12 Months
Arm/Group | Dasatinib, 100 mg | Imatinib, 800 mg
Started | 19 | 13
Completed | 11 | 3
Not Completed | 8 | 10
Not completed — Completed but did not enter extension | 5 | 3
Not completed — Sponsor terminated study | 2 | 2
Not completed — Lost to Follow-up | 0 | 1
Not completed — Enrollment failure | 0 | 1
Not completed — Adverse event unrelated to study drug | 1 | 0
Not completed — Investigator request | 0 | 1
Not completed — Study drug toxicity | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1
Period: Long-term (12-month) Extension
Arm/Group | Dasatinib, 100 mg | Imatinib, 800 mg
Started | 11 | 3
Completed | 2 | 1
Not Completed | 9 | 2
Not completed — Sponsor terminated study | 7 | 0
Not completed — Lack of major molecular response | 1 | 2
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dasatinib, 100 mg | Imatinib, 800 mg | Total
Number analyzed (Participants) | 19 | 13 | 32
Age, Customized [Mean (Standard Deviation); unit: Years] | 45.5 (14.83) | 53.2 (14.24) | 48.6 (14.85)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 3 | 9
  Male | 13 | 10 | 23
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 18 | 13 | 31
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Chronic Phase Chronic Myeloid Leukemia Who Have a Major Molecular Response (MMolR)
Description: MMolR is defined as reduction in transcript levels of the breakpoint cluster region (BCR)-V-abl Abelson murine leukemia viral oncogene homolog 1 (ABL) gene of at least 3 log. The BCR-ABL gene has a role in the production of a mutated protein that converts bone marrow stem cells from normal to leukemic.
Time Frame: At 12 months from baseline
Population: Efficacy analyses as originally described in the protocol were not conducted because of the low number of participants enrolled.
Arm/Group | Dasatinib, 100 mg | Imatinib, 800 mg
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Percentage of Participants With Death as Outcome, Adverse Events (AEs), Treatment-related AEs, Serious Adverse Events (SAEs), Treatment-related SAEs, and AEs Leading to Discontinuation
Description: AE=any new untoward medical occurrence or worsening of a preexisting medical condition that does not necessarily have a causal relationship with treatment. SAE=any untoward medical occurrence that at any dose results in death, persistent or significant disability/incapacity, drug dependency, or drug abuse; prolongs inpatient hospitalization; or is life-threatening, a congenital anomaly/birth defect, or an important medical event. Treatment related=possibly, probably, or certainly related to and of unknown relationship to study treatment.
Time Frame: Months 1 to 12, continuously, and Months 12 to 24, continuously
Population: All participants who received at least 1 dose of dasatinib or imatinib.
Measure: Number; unit: Percentage of participants
Arm/Group | Dasatinib, 100 mg | Imatinib, 800 mg
Number analyzed (Participants) | 19 | 13
Percentage of participants
  Deaths | 0 | 0
  AEs | 94.7 | 92.3
  Treatment-related AEs | 78.9 | 92.3
  SAEs | 15.8 | 7.7
  Treatment-related SAEs | 5.3 | 7.7
  AEs leading to discontinuation | 5.3 | 7.7

3. Secondary Outcome: Percentage of Participants With On-study AEs of Special Interest
Description: GI=gastrointestinal. AE=any new untoward medical occurrence or worsening of a preexisting medical condition that does not necessarily have a causal relationship with treatment. Grade 1=mild; Grade 2=moderate; Grade 3=severe and undesirable; Grade 4=life-threatening or disabling; Grade 5=death. Percentages based on the number of participants with a specific grade at baseline. Participants without on-study test values for a particular laboratory analyte are not included in the reporting of that analyte.
Time Frame: Months 1 to 12, continuously, and Months 12 to 24, continuously
Population: All participants who received at least 1 dose of dasatinib or imatinib.
Measure: Number; unit: Percentage of Participants
Arm/Group | Dasatinib, 100 mg | Imatinib, 800 mg
Number analyzed (Participants) | 19 | 13
Percentage of Participants
  Fluid retention (Any grade) | 5.3 | 38.5
  Fluid retention (Grades 3-5) | 0 | 7.7
  Fluid retention: Superficial edema (Any grade) | 0 | 30.8
  Fluid retention: Superficial edema (Grades 3-5) | 0 | 0
  Fluid retention: Generalized edema (Any grade) | 5.3 | 7.7
  Fluid retention: Generalized edema (Grades 3-5) | 0 | 7.7
  Hemorrhage (Any grade) | 0 | 15.4
  Hemorrhage (Grades 3-5) | 0 | 0
  Hemorrhage: GI bleeding (Any grade) | 0 | 7.7
  Hemorrhage: GI bleeding (Grades 3-5) | 0 | 0
  Hemorrhage: Other bleeding (Any grade) | 0 | 7.7
  Hemorrhage: Other bleeding (Grades 3-5) | 0 | 0
  Diarrhea (Any grade) | 26.3 | 30.8
  Diarrhea (Grades 3-5) | 0 | 0
  Skin rash (Any grade) | 42.1 | 15.4
  Skin rash (Grades 3-5) | 0 | 0

4. Secondary Outcome: Median Time to MMolR
Description: Time to MMolR is defined as the time from first treatment dose until measurement criteria are first met for MMolR. MMolR is defined as a reduction in transcript levels of the BCR-ABL gene of at least 3 log from baseline.
Time Frame: At 3, 6, 9, and 12 months from baseline
Population: as for outcome 1
Arm/Group | Dasatinib, 100 mg | Imatinib, 800 mg
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Percentage of Participants With Complete Cytogenetic Response
Description: Cytogenetic response is based on the prevalence of Ph+ metaphases among cells in metaphase in a bone marrow sample.
Time Frame: At 6 and 12 months from baseline
Population: as for outcome 1
Arm/Group | Dasatinib, 100 mg | Imatinib, 800 mg
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Median Time to Treatment Failure
Description: Time to treatment failure is defined as the time in days from randomization to progressive disease documented by the investigator, to death from any cause without prior progression, or to early treatment discontinuation for any reason, whichever occurs first. Participants without disease progression or who do not die and complete the 12-month study treatment are censored on the date of their last molecular, cytogenetic, or hematologic assessment.
Time Frame: Randomization to disease progression, death, or discontinuation (to 12 months)
Population: as for outcome 1
Arm/Group | Dasatinib, 100 mg | Imatinib, 800 mg
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Median Time to Progression-free Survival
Description: Progression-free survival is defined as the time in days from randomization to progressive disease documented by the investigator or to death from any cause without prior progression. Participants without progressive disease or who do not die and complete the 12-month treatment are censored on the date of their last molecular, cytogenetic, or hematologic assessment.
Time Frame: Randomization to disease progression or death (to 12 months)
Population: as for outcome 1
Arm/Group | Dasatinib, 100 mg | Imatinib, 800 mg
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Baseline to Month 12 and Month 12 to Month 24
Arm/Group | Dasatinib, 100 mg | Imatinib, 800 mg
Serious Adverse Events (participants affected / at risk) | 3/19 | 1/13
Other Adverse Events (participants affected / at risk) | 18/19 | 12/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dasatinib, 100 mg (N=19) | Imatinib, 800 mg (N=13)
MELAENA (Gastrointestinal disorders) | 0 | 1
HAEMATEMESIS (Gastrointestinal disorders) | 0 | 1
PNEUMONIA (Infections and infestations) | 1 | 0
SKIN BURNING SENSATION (Skin and subcutaneous tissue disorders) | 1 | 0
BREAST CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dasatinib, 100 mg (N=19) | Imatinib, 800 mg (N=13)
EYE PAIN (Eye disorders) | 1 | 0
EYE SWELLING (Eye disorders) | 0 | 1
EYE DISCHARGE (Eye disorders) | 1 | 0
EYELID OEDEMA (Eye disorders) | 0 | 1
CONJUNCTIVITIS (Eye disorders) | 0 | 2
EYE IRRITATION (Eye disorders) | 0 | 1
ORBITAL OEDEMA (Eye disorders) | 0 | 1
OCULAR HYPERAEMIA (Eye disorders) | 0 | 1
LACRIMATION INCREASED (Eye disorders) | 0 | 2
DACRYOSTENOSIS ACQUIRED (Eye disorders) | 1 | 0
BIOPSY (Investigations) | 1 | 0
CARDIAC MURMUR (Investigations) | 1 | 0
WEIGHT DECREASED (Investigations) | 1 | 0
BLOOD CALCIUM INCREASED (Investigations) | 1 | 0
BLOOD PHOSPHORUS DECREASED (Investigations) | 0 | 1
BLOOD PHOSPHORUS INCREASED (Investigations) | 1 | 0
ELECTROCARDIOGRAM QT INTERVAL (Investigations) | 0 | 1
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 2 | 0
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 2 | 0
BLOOD ALKALINE PHOSPHATASE INCREASED (Investigations) | 1 | 0
BLOOD LACTATE DEHYDROGENASE INCREASED (Investigations) | 1 | 0
ANGINA PECTORIS (Cardiac disorders) | 0 | 1
FLUSHING (Vascular disorders) | 0 | 1
HYPERTENSION (Vascular disorders) | 2 | 0
VENOUS INSUFFICIENCY (Vascular disorders) | 1 | 0
GOITRE (Endocrine disorders) | 0 | 1
ANXIETY (Psychiatric disorders) | 0 | 1
INSOMNIA (Psychiatric disorders) | 1 | 1
AGGRESSION (Psychiatric disorders) | 2 | 0
DEPRESSED MOOD (Psychiatric disorders) | 0 | 1
SEASONAL ALLERGY (Immune system disorders) | 1 | 0
HEADACHE (Nervous system disorders) | 8 | 4
MIGRAINE (Nervous system disorders) | 0 | 1
DIZZINESS (Nervous system disorders) | 1 | 0
DYSGEUSIA (Nervous system disorders) | 0 | 1
FACIAL PALSY (Nervous system disorders) | 0 | 1
FACIAL NEURALGIA (Nervous system disorders) | 0 | 1
DISTURBANCE IN ATTENTION (Nervous system disorders) | 0 | 1
NAUSEA (Gastrointestinal disorders) | 2 | 7
VOMITING (Gastrointestinal disorders) | 3 | 5
DIARRHOEA (Gastrointestinal disorders) | 5 | 4
DYSPEPSIA (Gastrointestinal disorders) | 1 | 1
TOOTHACHE (Gastrointestinal disorders) | 0 | 1
FLATULENCE (Gastrointestinal disorders) | 3 | 0
LIP BLISTER (Gastrointestinal disorders) | 1 | 0
CONSTIPATION (Gastrointestinal disorders) | 2 | 0
DENTAL CARIES (Gastrointestinal disorders) | 1 | 0
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 | 0
TOOTH DISORDER (Gastrointestinal disorders) | 1 | 0
ABDOMINAL DISCOMFORT (Gastrointestinal disorders) | 1 | 0
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 3 | 0
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 1 | 0
MALLORY-WEISS SYNDROME (Gastrointestinal disorders) | 0 | 1
GASTROINTESTINAL DISORDER (Gastrointestinal disorders) | 0 | 1
GASTROOESOPHAGEAL SPHINCTER INSUFFICIENCY (Gastrointestinal disorders) | 0 | 1
VERTIGO (Ear and labyrinth disorders) | 0 | 1
EAR PAIN (Ear and labyrinth disorders) | 0 | 1
TINNITUS (Ear and labyrinth disorders) | 2 | 0
INFECTION (Infections and infestations) | 0 | 1
INFLUENZA (Infections and infestations) | 1 | 0
SINUSITIS (Infections and infestations) | 1 | 1
BRONCHITIS (Infections and infestations) | 1 | 0
PHARYNGITIS (Infections and infestations) | 0 | 1
TONSILLITIS (Infections and infestations) | 1 | 0
EAR INFECTION (Infections and infestations) | 0 | 1
LABYRINTHITIS (Infections and infestations) | 1 | 0
ONYCHOMYCOSIS (Infections and infestations) | 1 | 1
GASTROENTERITIS (Infections and infestations) | 1 | 1
NASOPHARYNGITIS (Infections and infestations) | 2 | 2
TOOTH INFECTION (Infections and infestations) | 1 | 0
ORAL CANDIDIASIS (Infections and infestations) | 0 | 1
LOCALISED INFECTION (Infections and infestations) | 1 | 0
FUNGAL SKIN INFECTION (Infections and infestations) | 1 | 0
GASTROENTERITIS VIRAL (Infections and infestations) | 1 | 1
HERPES VIRUS INFECTION (Infections and infestations) | 0 | 1
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 | 0
DYSURIA (Renal and urinary disorders) | 0 | 1
NOCTURIA (Renal and urinary disorders) | 1 | 0
HAEMATURIA (Renal and urinary disorders) | 0 | 1
PROTEINURIA (Renal and urinary disorders) | 1 | 0
GOUT (Metabolism and nutrition disorders) | 1 | 0
HYPOKALAEMIA (Metabolism and nutrition disorders) | 1 | 0
FLUID RETENTION (Metabolism and nutrition disorders) | 1 | 0
DECREASED APPETITE (Metabolism and nutrition disorders) | 1 | 1
LYMPHOCYTOSIS (Blood and lymphatic system disorders) | 2 | 0
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 2 | 0
IRON DEFICIENCY ANAEMIA (Blood and lymphatic system disorders) | 1 | 0
RASH (Skin and subcutaneous tissue disorders) | 6 | 2
ECZEMA (Skin and subcutaneous tissue disorders) | 2 | 0
DRY SKIN (Skin and subcutaneous tissue disorders) | 1 | 1
PRURITUS (Skin and subcutaneous tissue disorders) | 2 | 0
URTICARIA (Skin and subcutaneous tissue disorders) | 1 | 0
SKIN ULCER (Skin and subcutaneous tissue disorders) | 1 | 0
RASH MACULAR (Skin and subcutaneous tissue disorders) | 1 | 0
RASH PAPULAR (Skin and subcutaneous tissue disorders) | 1 | 0
HYPERHIDROSIS (Skin and subcutaneous tissue disorders) | 1 | 0
RASH ERYTHEMATOUS (Skin and subcutaneous tissue disorders) | 0 | 1
PERIORBITAL OEDEMA (Skin and subcutaneous tissue disorders) | 0 | 2
DERMATITIS ACNEIFORM (Skin and subcutaneous tissue disorders) | 2 | 0
SKIN BURNING SENSATION (Skin and subcutaneous tissue disorders) | 1 | 0
BREAST MASS (Reproductive system and breast disorders) | 1 | 0
EPIDIDYMAL CYST (Reproductive system and breast disorders) | 1 | 0
TESTICULAR PAIN (Reproductive system and breast disorders) | 1 | 0
PRURITUS GENITAL (Reproductive system and breast disorders) | 1 | 0
THERMAL BURN (Injury, poisoning and procedural complications) | 1 | 0
MYALGIA (Musculoskeletal and connective tissue disorders) | 3 | 2
BACK PAIN (Musculoskeletal and connective tissue disorders) | 4 | 0
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 2 | 0
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 1 | 3
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 2 | 0
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 0 | 1
COUGH (Respiratory, thoracic and mediastinal disorders) | 3 | 1
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 1 | 1
DYSPHONIA (Respiratory, thoracic and mediastinal disorders) | 1 | 1
ORTHOPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 | 1
RHINORRHOEA (Respiratory, thoracic and mediastinal disorders) | 1 | 1
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 0 | 2
SPUTUM DISCOLOURED (Respiratory, thoracic and mediastinal disorders) | 0 | 2
INCREASED BRONCHIAL SECRETION (Respiratory, thoracic and mediastinal disorders) | 1 | 0
CHILLS (General disorders) | 1 | 0
OEDEMA (General disorders) | 0 | 1
FATIGUE (General disorders) | 7 | 3
MALAISE (General disorders) | 1 | 0
PYREXIA (General disorders) | 5 | 0
ASTHENIA (General disorders) | 1 | 3
CHEST PAIN (General disorders) | 1 | 1
FACIAL PAIN (General disorders) | 0 | 1
AXILLARY PAIN (General disorders) | 2 | 0
INFLUENZA LIKE ILLNESS (General disorders) | 3 | 0
MELANOCYTIC NAEVUS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0

LIMITATIONS AND CAVEATS:
Enrollment terminated prematurely on September 5, 2008, due to slow accrual. Only 32 of 156 planned participants were randomized from August 2, 2006. Per BMS standards, findings were reported in a synopsis format, with only safety results included.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication